CLINICAL TRIAL: NCT04988490
Title: Quantification of Endo- and Phytocannabinoids With Comparison to Pain Medication Requirements and Surgical Outcomes for Patients Undergoing Abdominal Surgery for Cancer
Brief Title: Quantification of Cannabinoids and Comparison to Post-Surgical Pain Medication Requirements and Surgical Outcomes
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Institute of Cannabis Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21-3544.cc; P30CA046934 (NIH); NCI-2021-08865 (Other: CTRP)
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Post-Surgical Pain; Post-Surgical Complication; Cancer; Cannabis Use
Keywords: Cannabis; Post-Surgical Complications; Post-Surgical Pain; Abdominal Surgery
MeSH Terms: conditions — Pain, Postoperative; Neoplasms; Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Daily cannabis users: Patients undergoing inpatient abdominal surgery for the treatment of cancer who self-report daily cannabis use
- Cannabis non-users: Patients undergoing inpatient abdominal surgery for the treatment of cancer who self-report no cannabis use

SUMMARY:
To determine how daily cannabis use affects surgical outcomes.

DETAILED DESCRIPTION:
To determine if patients who are daily cannabis users that are undergoing inpatient abdominal surgery for the treatment of cancer are different from non-cannabis users regarding phytocannabinoid and endocannabinoid levels, pain scores, pain medication requirements, and surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Undergoing abdominal surgery for the treatment of cancer
* Report no cannabis use in the last year or chronic cannabis use (defined as at least weekly use for 3 months or more)

Exclusion Criteria:

* patients with chronic pain, chronic pain syndrome on opioids
* female patients who are pregnant or lactating
* patients who report use of illicit substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients over the age of 18 undergoing inpatient abdominal surgery for the treatment of cancer who use cannabis daily prior to surgery or who are non-users of cannabis.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 30 days
  Postoperative opioid consumption among daily cannabis using and non-cannabis using patients undergoing abdominal surgery for cancer
Correlation of postoperative opioid consumption | 30 days
  Correlation between serum phytocannabinoid and endocannabinoid levels, pain scores, and postoperative opioid consumption
Correlation of postoperative complications | 30 days
  Correlation between 30-day post-operative complications, preoperative, and postoperative phytocannabinoid and endocannabinoid levels

CONTACTS AND LOCATIONS:
Overall Officials: Ana Gleisner, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided